CLINICAL TRIAL: NCT07214740
Title: A Phase 3B, Single-Arm, Open-Label, Multicenter Study to Evaluate the Safety of Pegcetacoplan in a Prefilled Syringe in Participants With Geographic Atrophy Secondary to Age-Related Macular Degeneration
Brief Title: Study to Evaluate a Pegcetacoplan (Syfovre®) Prefilled Syringe
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Apellis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APL2-GA-317
Record Dates: First submitted 2025-10-06; First posted 2025-10-09 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Geographic Atrophy Secondary to Age-related Macular Degeneration
Keywords: Geographic Atrophy; Age-Related Macular Degeneration
MeSH Terms: conditions — Geographic Atrophy; Macular Degeneration | interventions — pegcetacoplan

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pegcetacoplan, 15 mg/100 μL (single dose), intravitreal injection via prefilled syringe (Experimental): This is a 30-day, phase 3b, single-arm, open-label, multicenter study to evaluate the safety of IVT pegcetacoplan administered via PFS in participants with geographic atrophy (GA) secondary to age-related macular degeneration (AMD). The study consists of a screening/baseline visit at day 1, a follow-up call at day 7, and an end of study visit at day 30.
  Interventions: Drug: APL-2, Pegcetacoplan

INTERVENTIONS:
Drug: APL-2, Pegcetacoplan — Complement (C3) Inhibitor

SUMMARY:
This is a phase 3, open-label study to evaluate the safety of pegcetacoplan in a prefilled syringe (PFS)

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be aged at least 60 years and have a diagnosis of GA secondary to AMD.
2. Participants must have adequate clarity of ocular media, adequate pupillary dilation, and fixation to permit the collection of good quality images in the study eye as determined by the retina specialist.
3. Study eye must be deemed to be indicated for IVT pegcetacoplan therapy at the discretion of the retina specialist.
4. Female participants must be women of nonchildbearing potential, defined as postmenopausal women with 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (eg, age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy, or tubal ligation at least 6 weeks prior to screening/baseline. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow-up hormone level assessment is she considered not of childbearing potential.
5. Male participants must be surgically sterile or must agree to use protocol-defined highly effective methods of contraception and to refrain from donating sperm from screening through the duration of the study and for 90 days after their dose of study drug.
6. Participants must be willing and able to provide informed consent and comply with the study visit schedule and study-related procedures/requirements.

Exclusion Criteria:

1. Retinal atrophy secondary to a condition other than AMD, such as Stargardt disease, cone rod dystrophy, or toxic maculopathies like plaquenil maculopathy, in either eye.
2. Any history or active CNV associated with AMD or any other cause, including any evidence of RPE rips or evidence of neovascularization anywhere based on spectral domain optical coherence tomography imaging as assessed by the retina specialist.
3. Presence of an active ocular disease in the study eye that, in the opinion of the investigator, compromises or confounds visual function, including but not limited to, uveitis and other macular diseases (eg, clinically significant epiretinal membrane, full thickness macular hole, or uncontrolled glaucoma/ocular hypertension); benign conditions in the opinion of the investigator, such as peripheral retina dystrophy, are not exclusionary.
4. IOP >21 mm Hg in the study eye at the screening/baseline visit.
5. Participants who have legal blindness or worse vision in study eye (ie, best-corrected visual acuity [BCVA] of ≤35 Early Treatment Diabetic Retinopathy Study letters).
6. History of laser therapy in the macular region of study eye.
7. Any intraocular surgery in the study eye at any time during the past 3 months.
8. Any ocular condition other than GA secondary to AMD that may require surgery or medical intervention during the study period or, in the opinion of the investigator, could compromise visual function during the study period.
9. Any prior extended-release therapeutic agent, or ocular drug-release device implantation (approved or investigational, including steroids) in the study eye.
10. Active, suspected, or history of IOI in either eye at the screening/baseline visit.
11. Any contraindication to IVT injection, including current ocular or periocular infection.
12. Current systemic infectious disease or a therapy for active infectious disease.
13. History of IVT injection in the study eye within 90 days or 5 half-lives of the product (other than IVT pegcetacoplan), whichever is longer, prior to the screening/baseline visit
14. Participation in an investigational product or medical device study (other than IVT pegcetacoplan studies) within 90 days or 5 half-lives of the product, whichever is longer, prior to the screening/baseline visit.
15. Known hypersensitivity to pegcetacoplan or any of the excipients in pegcetacoplan solution.
16. Pregnancy or breastfeeding

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2025-10-24 (Actual); Primary Completion 2025-12-12 (Actual); Study Completion 2025-12-12 (Actual)

PRIMARY OUTCOMES:
To evaluate safety and tolerability of intravitreal (IVT) pegcetacoplan administered via PFS by assessing incidence of ocular treatment-emergent adverse events (TEAEs) in the study eye | Up to Day 30

SECONDARY OUTCOMES:
The number of IVT pegcetacoplan injections successfully administered using PFS as reported by retina specialists immediately following the injection | At Day 1

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - California Retina Consultants, Bakersfield, California
  - California Retina Consultants, Oxnard, California
  - Austin Retina Associates, Austin, Texas
  - Retina Consultants of Texas, Katy, Texas
  - Retina Consultants of Texas, Woodland, Texas